CLINICAL TRIAL: NCT05461417
Title: Non-comparative Prospective Study Evaluating the Long-term Efficacy, Tolerance and Compliance of the Panthera D-SAD Mandibular Advancement Orthosis in the Management of Obstructive Sleep Apnea Hypopnea Syndrome (PANTHERA Study)
Brief Title: Long-term Efficacy, Tolerance and Compliance of Panthera D-SAD® Mandibular Advancement Orthosis in Sleep Apnea
Acronym: PANTHERA
Status: Active, not recruiting | Type: Observational
Sponsor: Panthera Dental Inc. (Industry)
Collaborators: AXONAL (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRO-140
Record Dates: First submitted 2022-06-29; First posted 2022-07-18 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea Hypopnea Syndrome (OSAS); snoring; Mandibular Advancement Orthosis; Panthera D-SAD
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- D-SAD group: Patients equipped with Panthera D-SAD MAO
  Interventions: Device: D-SAD

INTERVENTIONS:
Device: D-SAD — Patients equipped with Panthera D-SAD® orthosis will be recruited.

SUMMARY:
Obstructive sleep apnea (OSA) is a common, chronic and serious medical condition. Oral appliance therapy (OAT) also called mandibular advancement orthosis (MAO) provides long-term therapy for OSA patients. The Panthera D-SAD® is a computer aided design (CAD)/computer aided manufacturing (CAM), patient-matched, 3D printed, biocompatible nylon OAT. This five-year, observational prospective and multicenter study will assess the effectiveness of the PANTHERA D-SAD® orthosis on reducing the apnea hypopnea index (AHI) and obstructive sleep apnea-hypopnea syndrome (OSAHS) symptoms. Adherence, tolerance, and side effects will be evaluated.

An estimated ten sites composed of a professional dyad, a specialist in sleep disorders, and a practitioner with knowledge of both sleep and the manducatory apparatus will recruit 337 patients. The entry criteria include an AHI between 15 and 30 or higher if the patient meets certain medical and dental criteria, no prior use of OAT, and struggles or refuses continuous positive airway (CPAP) treatment. The professional collaborative nature of the study reflects real-world clinical practice.

Participants will be followed over the course of five years at the following time points. Visits include the following: Specialist in sleep disorders: (1) Inclusion, (2) 3 months, (3) 2 years, (4) 5 years. Specialist in manducatory apparatus (dentist): (1) Inclusion, orthosis set-up and titration, (2) 6 months, (3) 2 and (4) 5 years The efficacy of the Panthera D-SAD® MAO will be assessed by the treatment success rate at five years, defined as a reduction ≥ 50% in the initial AHI, when monitored by nocturnal breathing polygraphy (NP) or polysomnography (PSG). Secondary endpoints will also be obtained at the aforementioned time points for reporting. The results of this study will fulfill regulatory requirements for reimbursement in France.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18
* Moderate OSAHS or severe OSAHS and refuse or intolerance to treatment with continuous positive pressure
* Patient who has never worn MAO
* Accepting and able to complete questionnaires in French on the impact of their disease and their quality of life
* Informed and having signed a written consent
* Affiliated to a social security system

Exclusion Criteria:

* One or more contraindications to wearing a mandibular advancement orthosis
* Central sleep apnea
* Severe OSAHS associated with another sleep pathology
* Serious respiratory disorders other than OSAS
* Severe psychiatric or neurological disorders
* Progressive cancer and/or chronic joint, inflammatory or immunosuppressive disease
* Known allergy to one of the components of the medical device
* Simultaneous participation in another intervention research
* Vulnerable subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from moderate sleep apnea, or severe sleep apnea with refusal or failure of CPAP treatment and meeting the eligibility criteria may participate in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the MAO Panthera D-SAD® evaluated by the success rate of the treatment at 5 years | At 5 years after treatment start
  Proportion of patients with a reduction in AHI of 50% or more compared to inclusion, measured by polygraphy or somnopolygraphy

SECONDARY OUTCOMES:
AHI evolution according to severity | Inclusion, 3 months, 2 years, 5 years
  AHI mean in global and in severity subgroups
Change in AHI | 3 months, 2 years, 5 years
  Difference between AHI at visit and at baseline
Description of severity groups | Inclusion, 3 months, 2 years, 5 years
  Proportion of patients with AHI ≤ 5, ≤ 15 and ≤ 30 at visit
Description of tiredness | Inclusion, 3 months, 2 years, 5 years
  Mean score of Pichot scale at each visit
Description of sleepiness | Inclusion, 3 months, 2 years, 5 years
  Mean score of Epworth scale at each visit
Description of snoring | Inclusion, 3 months, 2 years, 5 years
  Mean score of snoring measured by a Likert scale at each visit
Quality of life assessed by Nottingham Health Profile (NHP) questionnaire | 3 months, 2 years, 5 years
  Mean score of Nottingham Health Profile (NHP) at each visit
Satisfaction assessed by a Likert scale | 3 months, 2 years, 5 years
  Mean score of satisfaction measured by a Likert scale at each visit
Oxygen Desaturation Index (ODI) evolution | 3 months, 2 years, 5 years
  Difference between ODI at visit and at baseline
Minimal oxygen saturation (SpO2) | Inclusion, 3 months, 2 years, 5 years
  Minimum Spo2 at visit
Duration with SpO2<90% | Inclusion, 3 months, 2 years, 5 years
  Duration with SpO2<90%
Observance | Inclusion, 3 months, 2 years, 5 year
  Number of nights equipped for a week, number of hours equipped for a night, percentage of patients equipped ≥4h per night
Dental tolerance | Inclusion, during titration, at 3 and 6 months then at 1, 2, 3, 4, 5 years
  Number of device adverse reaction (DAR), proportion of patients with at least one DAR, number of incidents and deficiencies
Titration description | during titration
  Rod length corresponding to optimal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GAGNADOUX, Prof, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No